CLINICAL TRIAL: NCT05427864
Title: Comparison of Multiparametric Prostate MRI and Ga-68 PSMA PET Imaging in Prostate Cancer Staging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Can Sicimli, Principal Investigator, Gulhane Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GULHANEUROCANSICIMLI001
Record Dates: First submitted 2022-06-11; First posted 2022-06-22 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Prostate Cancer; Prostate Cancer Stage
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: 47 male patients who will be evaluated with both imaging studies will be included in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Multiparametric Prostate MRI — Comparison of Ga68 PSMA PET and Multiparametric Prostate MR imaging tests used in staging in patients diagnosed with prostate cancer
  Other Names: Ga-68 PSMA PET

SUMMARY:
In this study, it is aimed to compare the lesion location, lesion size, local and distant metastases detection rates of Ga68 PSMA PET and Multiparametric Prostate MR imaging tests used in staging in patients diagnosed with prostate cancer.

The pathologies of the patients who were decided to undergo radical prostatectomy as a treatment will also be compared with the staging tests.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with prostate cancer
* Gleason score 7 or above / 6 with high risk
* No other treatment

Exclusion Criteria:

* treated with radiotherapy
* treated with ADT

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Because of prostate cancer study
Enrollment: 47 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-01-05 (Estimated); Study Completion 2023-03-05 (Estimated)

PRIMARY OUTCOMES:
Lesion location | Between prostate biopsy and curative treatment decision , usually 2 month
  Both MRI and PET results will be compared. Lesion location will be defined as "left", "right", "apical", "basal", "midline".
Lesion Size | Between prostate biopsy and curative treatment decision , usually 2 month
  Both MRI and PET results will be compared, Lesion size will be stated in milimeters.
Lymph node involvement | Between prostate biopsy and curative treatment decision , usually 2 month
  Both MRI and PET results will be compared. Involvement will be stated as "exist", "non-exist".
Extraprostatic involvement | Between prostate biopsy and curative treatment decision , usually 2 month
  Both MRI and PET results will be compared. Involvement will be stated as "exist" , "non-exist".
Local and distant metastasis | Between prostate biopsy and curative treatment decision , usually 2 month
  Both MRI and PET results will be compared. Metastasis will be stated as "exist" , "non-exist".

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane Research and Training Hospital, Ankara, Etlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided